CLINICAL TRIAL: NCT05791708
Title: Cold Agglutinin Disease Real World Evidence Registry
Acronym: CADENCE
Status: Recruiting | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS16454; EUPAS47940 (Registry Identifier: ENCePP); U1111-1287-7090 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-02-15; First posted 2023-03-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cold Agglutinin Disease (CAD); Cold Agglutinin Syndrome (CAS)
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — sutimlimab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cold agglutinin disease (CAD): Patient with a diagnosis of CAD as per investigator judgment based on the diagnosis criteria listed in study protocol. In addition, this group includes a cohort of CAD patients treated with sutimlimab
  Interventions: Drug: Sutimlimab
- cold agglutinin syndrome (CAS): Patient with a diagnosis of CAS as per investigator judgment based on the diagnosis criteria listed in study protocol

INTERVENTIONS:
Drug: Sutimlimab — CAD patients in Sutimlimab cohort must be treated according to routine clinical practice
  Groups: cold agglutinin disease (CAD)

SUMMARY:
This is a multinational, multi-center, observational, prospective, longitudinal disease registry designed to collect data on participants with cold agglutinin disease (CAD) or cold agglutinin syndrome (CAS). Among them, a minimum of 30 patients with CAD treated with sutimlimab are expected to take part in the sutimlimab cohort study. Patients with CAD who have been enrolled in previous sutimlimab clinical trials (e.g., BIVV009-01/LTS16214 [NCT02502903,CAD patients], BIVV009-03/EFC16215 [NCT03347396], and BIVV009-04/EFC16216 [NCT03347422]) and who either completed or discontinued the corresponding clinical trial are eligible to participate in the registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥18 years
2. Patient able to understand the purpose of the study and who (or whose legally authorized representative) provided signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations
3. Patient with a diagnosis of CAD or CAS as per Investigator judgment based on the diagnosis criteria listed in study protocol

Exclusion Criteria:

1. Patient with mixed warm and cold autoimmune hemolytic anemia, or warm autoimmune hemolytic anemia
2. Patient actively participating in a CAD or CAS interventional clinical trial. After a patient completes participation in said trial, he/she may be eligible for enrollment in this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with CAD or CAS will be eligible, regardless of the type of CAD or CAS-specific therapy they are receiving. In addition, the Cadence registry will include a sutimlimab cohort study whose objective is to assess the safety and the effectiveness of sutimlimab in patients with CAD in a real-world setting.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2028-11-02 (Estimated); Study Completion 2028-11-02 (Estimated)

PRIMARY OUTCOMES:
Patterns of CAD and CAS disease characteristics | Up to 6 years
  CAD or CAS characteristics at diagnosis, enrollment, and during follow up (e.g., criteria used for diagnosis, symptoms, laboratory results) will be described.
Number of participants with CAD or CAS complications | Up to 6 years
  Thromboembolic events (venous, arterial or cerebral), deaths related to CAD or CAS, other CAD/CAS complications (e.g., acute hemolytic crisis, hemolysis-related complications), and other comorbid conditions occurring before enrollment, at enrollment, and during follow up will be described.
Patterns of use of CAD and CAS treatments | Up to 6 years
  CAD or CAS treatments received before enrollment, at enrollment, and during the follow up period will be summarized. CAD or CAS symptoms and complications, autoimmune disorders or lymphoproliferative disorders, physician assessment of treatment status, and changes in laboratory results will be described by CAD or CAS treatments.
Number of participants with health-resource utilization | Up to 6 years
  Health resource utilization may include hospitalizations (including length of stay), outpatient visits, emergency room visits, specific transfusion visits, nursing home/rehabilitation center stays, and home healthcare visits during registry follow-up period
Cold Agglutinin Disease Symptoms and Impact Questionnaire (CAD-SIQ) | Up to 6 years
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Up to 6 years
36-Item Short Form Survey Instrument (SF-36) v2 | Up to 6 years
Sutimlimab cohort: Sutimlimab treatment patterns | Up to 6 years
  Sutimlimab dosing information, reasons for dose adjustments, reasons for discontinuation will be described.
Sutimlimab cohort: Number of participants with adverse events, serious adverse events, adverse events of special interests (AESIs), other events of interests (e.g., Treatment emergent) | Up to 6 years
Sutimlimab cohort: change from baseline in hemoglobin | From baseline up to 6 years
Sutimlimab cohort: change from baseline in bilirubin | From baseline up to 6 years
Sutimlimab cohort: change from baseline in Lactate dehydrogenase (LDH) | From baseline up to 6 years
Sutimlimab cohort: number of blood cells transfusions | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Alvarez Rojo, Study Director — RECORDATI GROUP
Locations (68):
- United States (19):
  - University of Alabama at Birmingham Site Number : 1230, Birmingham, Alabama
  - SLO Oncology and Hematology Site Number : 1235, San Luis Obispo, California
  - Mission Hope Medical Oncology Site Number : 1241, Santa Maria, California
  - MedStar Georgetown University Hospital / Lombardi Comprehensive Cancer Center Site Number : 1208, Washington D.C., District of Columbia
  - Piedmont Cancer Institute, P.C Site Number : 1226, Atlanta, Georgia
  - Orchard Heathcare Research Inc. Site Number : 1202, Skokie, Illinois
  - Siouxland Regional Cancer Center dba June E. Nylen Cancer Center Site Number : 1220, Sioux City, Iowa
  - Reliant Medical Group Site Number : 1205, Worcester, Massachusetts
  - Henry Ford Hospital Site Number : 1232, Detroit, Michigan
  - Northwell Health-Monter Cancer Center-North Shore University Hospital and Steven and Alexandra Cohen Children's Medical Center of New York (Schneider Children's Hospital)-North Shore Long Island Jewis Site Number : 1231, Lake Success, New York
  - Center for Blood Disorders Site Number : 1214, New York, New York
  - SUNY Upstate Medical University Site Number : 1221, Syracuse, New York
  - Brody School of Medicine at East Carolina University Site Number : 1203, Greenville, North Carolina
  - Cleveland Clinic Foundation Site Number : 1207, Cleveland, Ohio
  - The Ohio State University Site Number : 1236, Columbus, Ohio
  - Hematology Oncology Associates, PC Site Number : 1211, Medford, Oregon
  - University of Pittsburgh Medical Center-UPMC Hillman Cancer Center Site Number : 1210, Pittsburgh, Pennsylvania
  - UT Medical Center Cancer Institute Site Number : 1237, Knoxville, Tennessee
  - University of Washingtion Seattle Cancer Care Alliance Site Number : 1238, Seattle, Washington
- Austria (2):
  - Investigational Site Number : 3101, Salzburg
  - Investigational Site Number : 3102, Vienna
- France (16):
  - Investigational Site Number : 3222, Amiens
  - Investigational Site Number : 3214, Angers
  - Investigational Site Number : 3204, Cesson-Sévigné
  - Investigational Site Number : 3211, Chalon-sur-Saône
  - Investigational Site Number : 3206, Corbeil-Essonnes
  - Investigational Site Number : 3201, Créteil
  - Investigational Site Number : 3219, Dijon
  - Investigational Site Number : 3221, Epagny-Metz-Tessy
  - Investigational Site Number : 3217, Paris
  - Investigational Site Number : 3213, Pau
  - Investigational Site Number : 3203, Pessac
  - Investigational Site Number : 3216, Poitiers
  - Investigational Site Number : 3202, Quimper
  - Investigational Site Number : 3220, Rennes
  - Investigational Site Number : 3205, Saint-Priest-en-Jarez
  - Investigational Site Number : 3218, Toulouse
- Germany (3):
  - Investigational Site Number : 3301, Essen
  - Investigational Site Number : 3306, Hanover
  - Investigational Site Number : 3302, Landshut
- Italy (9):
  - Investigational Site Number : 3413, Brescia, Lombardy
  - Investigational Site Number : 3410, Campobasso
  - Investigational Site Number : 3403, Novara
  - Investigational Site Number : 3411, Palermo
  - Investigational Site Number : 3415, Pavia
  - Investigational Site Number : 3412, Ravenna
  - Investigational Site Number : 3402, Reggio Calabria
  - Investigational Site Number : 3404, Roma
  - Investigational Site Number : 3405, Terni
- Japan (2):
  - Investigational Site Number : 2203, Fukushima, Fukushima
  - Investigational Site Number : 2204, Himeji-shi, Hyōgo
- Spain (2):
  - Investigational Site Number : 3701, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 3712, Madrid
- United Kingdom (15):
  - Investigational Site Number : 3603, Truro, Cornwall
  - Investigational Site Number : 3617, Carlisle, Cumbria
  - Investigational Site Number : 3608, Gillingham, Kent
  - Investigational Site Number : 3605, London, London, City of
  - Investigational Site Number : 3602, Salford, Manchester
  - Investigational Site Number : 3623, Airdrie, North Lanarkshire
  - Investigational Site Number : 3601, Newcastle upon Tyne, North Tyneside
  - Investigational Site Number : 3613, Middlesbrough, North Yorkshire
  - Investigational Site Number : 3611, Oxford, Oxfordshire
  - Investigational Site Number : 3606, Taunton, Somerset
  - Investigational Site Number : 3618, Birmingham
  - Investigational Site Number : 3620, Harrow
  - Investigational Site Number : 3612, Leeds
  - Investigational Site Number : 3607, Liverpool
  - Investigational Site Number : 3621, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.